CLINICAL TRIAL: NCT02547129
Title: A Randomized Clinical Trial of Static Versus Articulating Antibiotic Spacer for Treatment of Periprosthetic Joint Infection in Total Knee Arthroplasty
Brief Title: Static vs. Articulating Antibiotic Spacer for Periprosthetic Joint Infection in Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling patients as patients wanted articulating spacers.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael J. Taunton, M.D., Assistant Professor of Orthopedics, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-003291
Record Dates: First submitted 2015-08-18; First posted 2015-09-11 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Prosthetic Joint Infection of the Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Static Antibiotic Spacer (Active Comparator): Patient with prosthetic joint infection of their knee will have a two stage joint replacement surgery with the Static Antibiotic Spacer Surgical Implant being used to treat the joint infection until the second stage of surgery which will replace the joint after the infection is treated.
  Interventions: Device: Static Antibiotic Spacer Surgical Implant
- Articulating Antibiotic Spacer (Active Comparator): Patient with prosthetic joint infection of their knee will have a two stage joint replacement surgery with the Articulating Antibiotic Spacer Surgical Implant being used to treat the joint infection until the second stage of surgery which will replace the joint after the infection is treated.
  Interventions: Device: Articulating Antibiotic Spacer Surgical Implant

INTERVENTIONS:
Device: Static Antibiotic Spacer Surgical Implant — Joint spacer for treatment of joint infection
  Arms: Static Antibiotic Spacer
Device: Articulating Antibiotic Spacer Surgical Implant — Joint spacer for treatment of joint infection
  Arms: Articulating Antibiotic Spacer

SUMMARY:
The primary aim of the study is to compare two techniques for treatment of total knee infection: resection total knee arthroplasty with an articulating (motion in the joint) spacer and resection total knee arthroplasty with a static (no motion in the joint) spacer.

ELIGIBILITY:
Inclusion Criteria

1. Male or female age 18 to 100 years of age.
2. Preoperative diagnosis of bacterial infection by culture which would include a preoperative aspiration and at least three intraoperative cultures. The preoperative aspiration would also be sent for a cell count with differential. All patients would have an erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP) drawn in the preoperative phase. Patients with a negative preoperative aspiration, but an actively draining wound or draining sinus tract, would be considered as infected. Intraoperative histopathology would also be obtained in all cases of infected total knee replacement at the time of the resection.
3. Intact extensor mechanism.
4. Adequate soft tissue envelope (no requirement for soft tissue coverage such as a muscle flap or skin graft)
5. Adequate bone stock for knee reconstruction
6. Medical fitness for staged knee reconstruction

Exclusion Criteria

1. Known Atypical infection (mycobacterial or fungal)
2. Extensor mechanism disruption
3. Inadequate soft tissue envelope requiring muscle flap or skin grafting
4. Inadequate bone stock (T3 or F3 by the Anderson Orthopaedic Research Institute (AORI) classification)
5. Medical status precluding staged knee reconstruction
6. Requirement for hinged knee reconstruction at the time of reimplantation
7. Pregnant women - for women of child bearing age, a negative pregnancy test will be needed prior to enrollment to the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01-23 (Actual); Study Completion 2017-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Taunton, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Static Antibiotic Spacer | Articulating Antibiotic Spacer
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Difficulty with ongoing infection | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Static Antibiotic Spacer | Articulating Antibiotic Spacer | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Non-Hispanic or Latino | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Repeat Infections
Description: The rate of repeat infections after re-implantation Total Knee Arthroplasty.
Time Frame: 1 year post-operatively
Population: Study was terminated early due to difficulty enrolling patients.
Arm/Group | Static Antibiotic Spacer | Articulating Antibiotic Spacer
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Total Knee Replacement Functional Scores
Description: Functional scores were measured using the Knee Society Score, a clinical standard for rating the outcome of total knee replacements. Scores range from 0 -100, where a higher score reflects a more positive outcome for the subject.
Time Frame: baseline, 1 year post-operatively
Population: Study was terminated early due to difficulty enrolling patients.
Arm/Group | Static Antibiotic Spacer | Articulating Antibiotic Spacer
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pre-operative Range of Motion (ROM)
Description: The degree of knee flexion was measured pre-operatively.
Time Frame: baseline
Population: Study was terminated early due to difficulty enrolling patients.
Arm/Group | Static Antibiotic Spacer | Articulating Antibiotic Spacer
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Post-operative Range of Motion (ROM)
Description: The degree of knee flexion was measured one year post-operatively.
Time Frame: 1 year post-operatively
Population: Study was terminated early due to difficulty enrolling patients.
Arm/Group | Static Antibiotic Spacer | Articulating Antibiotic Spacer
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Static Antibiotic Spacer | Articulating Antibiotic Spacer
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
The study was terminated early due to difficulty in enrolling patients, as patients wanted articulating spacers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT02547129/Prot_SAP_000.pdf